CLINICAL TRIAL: NCT03689595
Title: Predicting Progression of Developing Myeloma in a High-Risk Screened Population (PROMISE)
Status: Recruiting | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Irene Ghobrial, MD, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 18-370
Record Dates: First submitted 2018-09-20; First posted 2018-09-28 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We collect blood samples from participants to test for precursor conditions to multiple myeloma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Specimen Collection: * Samples of blood (2-4 tablespoons) from 4 tubes will be collected
  * Analysis will be performed on the blood to test for multiple myeloma precursor conditions.
  Interventions: Other: Sample of Blood

INTERVENTIONS:
Other: Sample of Blood — Collection of blood sample from participants

SUMMARY:
The PROMISE Study aims to establish a prospective cohort of individuals with precursor conditions to multiple myeloma, such as monoclonal gammopathy of undetermined significance (MGUS) and smoldering multiple myeloma (SMM). We will study these patients as a means to identify risk factors for progression to symptomatic multiple myeloma.

DETAILED DESCRIPTION:
The goal of the PROMISE research study is to determine clinical/genomic alterations present in individuals with MGUS and SMM, who are diagnosed through screening of a high-risk population. We also seek to determine clinical/genomic/epigenetic and immune environmental predictors of progression to multiple myeloma in patients with MGUS and SMM.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 30 years
* AA race (self-identified) and/or first-degree relative of a patient with a plasma cell dyscrasia such as MGUS, SMM, MM, and Waldenström's Macroglobulinemia, or another blood cancer.
* Those over 18 are also eligible if they have 2 or more family members with a blood cancer

Exclusion Criteria:

* • Persons diagnosed with cancer at any site (including hematologic cancers) with symptomatic disease requiring active therapy.

• Persons with an already diagnosed plasma cell dyscrasia such as MGUS, SMM, MM, and Waldenström's Macroglobulinemia

First-degree relatives would not need to be identified by the participant.

This study includes all special populations who fall within the eligible high-risk age range, ≥ 30 years of age, including adults unable to consent, pregnant women, and prisoners. These populations will not be excluded as this is a non-therapeutic study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All special populations who fall within the eligible high-risk age range, ≥ 30 years of age are included.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2018-10-31 (Actual); Primary Completion 2033-10-31 (Estimated); Study Completion 2033-10-31 (Estimated)

PRIMARY OUTCOMES:
Time to progression (TTP) from MGUS/SMM to overt multiple myeloma. | 15 years
  Progression to symptomatic multiple myeloma

CONTACTS AND LOCATIONS:
Overall Officials: Irene Ghobrial, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bertamini L, Alberge JB, Lee DJ, El-Khoury H, Kim S, Fleming G, Murphy C, Colchie J, Davis MI, Perry J, Lightbody ED, Allam S, Goqwana LN, Philip V, Smyth N, Sakrikar D, Perkins M, Harding S, Troske D, Getz G, Karlson EW, Munshi N, Anderson KC, Trippa L, Marinac CR, Chen WC, Joffe M, Ghobrial IM. Serum free light chains in a racially diverse population including African Americans and populations from South Africa. Blood. 2025 Feb 20;145(8):840-849. doi: 10.1182/blood.2024026078. PMID 39571144
- [Derived] Lee DJ, El-Khoury H, Tramontano AC, Alberge JB, Perry J, Davis MI, Horowitz E, Redd R, Sakrikar D, Barnidge D, Perkins MC, Harding S, Mucci L, Rebbeck TR, Ghobrial IM, Marinac CR. Mass spectrometry-detected MGUS is associated with obesity and other novel modifiable risk factors in a high-risk population. Blood Adv. 2024 Apr 9;8(7):1737-1746. doi: 10.1182/bloodadvances.2023010843. PMID 38212245
- [Derived] El-Khoury H, Lee DJ, Alberge JB, Redd R, Cea-Curry CJ, Perry J, Barr H, Murphy C, Sakrikar D, Barnidge D, Bustoros M, Leblebjian H, Cowan A, Davis MI, Amstutz J, Boehner CJ, Lightbody ED, Sklavenitis-Pistofidis R, Perkins MC, Harding S, Mo CC, Kapoor P, Mikhael J, Borrello IM, Fonseca R, Weiss ST, Karlson E, Trippa L, Rebbeck TR, Getz G, Marinac CR, Ghobrial IM. Prevalence of monoclonal gammopathies and clinical outcomes in a high-risk US population screened by mass spectrometry: a multicentre cohort study. Lancet Haematol. 2022 May;9(5):e340-e349. doi: 10.1016/S2352-3026(22)00069-2. Epub 2022 Mar 25. PMID 35344689